CLINICAL TRIAL: NCT06842563
Title: A Multicenter Clinical Trial to Evaluate the Clinical Performance and Accuracy of the Human DAB2IP, CHFR, and GRASP Gene Methylation Kit (PCR-fluorescence Probe) in Patients With Suspected Hepatocellular Carcinoma
Brief Title: Hepatocellular Carcinoma 3 Gene Methylation Combination Detection Kit (PCR Fluorescent Probe Method) Multicenter Clinical Trial
Status: Active, not recruiting | Type: Observational
Sponsor: Singlera Genomics Inc. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SGI-PCR-02
Record Dates: First submitted 2025-02-13; First posted 2025-02-24 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular carcinoma; HBV or HCV infection; Nonalcoholic steatohepatitis; Liver cirrhosis; Benign hepatopathy; Family history of liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B; Hepatitis C; Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma sample DNA sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (2):
- Case group: Hepatocellular carcinoma (including stage I-IV) for initial treatment
- control group: Hepatitis, cirrhosis, benign lesions of the liver and other tumors (esophageal, gastric, bile duct, bowel, breast, lung, pancreatic, prostate cancer)

SUMMARY:
This clinical trial aims to systematically evaluate the clinical performance and accuracy of the HepaAiQ test kit, a multi-gene methylation assay based on PCR with fluorescent probe detection. The test results are compared against clinical reference standards, including pathological and/or imaging diagnoses, to assess the product's diagnostic performance. Additionally, for each gene detectable by the HepaAiQ assay, digital PCR is used as a comparator to validate analytical accuracy. The dual approach-clinical and analytical validation-supports the intended use of the test and provides sufficient clinical evidence for its registration and regulatory submission in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, gender unlimited;
2. Subjects for whom sufficient blood samples can be obtained (whole blood volume not less than 10 mL);
3. The performance of the blood-based, multi-gene methylation test is being evaluated in a diverse population including:

   (i) Treatment-naïve individuals presenting with signs and/or symptoms suggestive of hepatocellular carcinoma (HCC) as assessed by clinicians; (ii) Individuals at high risk for liver cancer, including those with HBV or HCV infection, excessive alcohol intake, non-alcoholic steatohepatitis (NASH), liver cirrhosis of various etiologies (LC), benign hepatic lesions (BHL), or a family history of liver cancer; (iii) Patients with other malignancies, including but not limited to esophageal, gastric, colorectal, pancreatic, lung, breast, and prostate cancers.
4. Voluntarily participate in the experiment and sign the informed consent.

Exclusion Criteria:

1. Liver cancer subjects who have received previous treatment, such as radiotherapy and chemotherapy, surgery, etc.;
2. Subjects with other malignant tumors;
3. Subjects with recurrent liver cancer confirmed or suspected by the investigator;
4. Subjects whose information is missing or untraceable;
5. The researcher believes that the subjects should not be included in this study for other reasons.

Min Age: 18 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: (i) Initial treatment subjects with symptoms and/or signs suspected of hepatocellular carcinoma as determined by the clinician;
  People with HBV or HCV infection, excessive alcohol consumption, non-alcoholic steatohepatitis, cirrhosis of the liver from other causes (LC), benign hepatopathy (BHL), and a family history of liver cancer;
  iii Subjects with other tumors, including but not limited to esophageal, stomach, colorectal, pancreatic, lung, breast, prostate, etc
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Study on the clinical performance of human DAB2IP, CHFR and GRASP gene methylation detection kit (PCR-fluorescent probe method) | From enrollment to the end of detection at 16 week
  By comparing the test reagent with the clinical reference standard (pathological diagnosis and/or imaging diagnosis), the test results of the test reagent were compared with the clinical reference standard to verify the clinical performance of the product

SECONDARY OUTCOMES:
Accuracy of human DAB2IP, CHFR and GRASP gene methylation detection kit (PCR-fluorescent probe method) | From enrollment to the end of detection at 16 week
  For each gene detected by the test reagent, the digital PCR method was used as a comparison method to verify the accuracy of the test reagent detection

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University in Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial